CLINICAL TRIAL: NCT05476913
Title: A Randomised Controlled Trial of the Effectiveness of Intermittent Surface Neuromuscular Stimulation Using the Geko™ Device Compared With Intermittent Pneumatic Compression to Prevent Venous Thromboembolism in Immobile Acute Stroke Patients
Brief Title: GEKO Venous Thromboembolism Prevention Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Keele University (Other); University Hospitals of North Midlands NHS Trust (Other); University of California (Other); Bournemouth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FSK-VTE-001; ISRCTN11175235 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2022-07-21; First posted 2022-07-27 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Acute; Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: geko; intermittent pneumatic compression; Stroke, Acute; Venous Thromboembolism; Pulmonary Embolism; DVT prophylaxis
MeSH Terms: conditions — Stroke; Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: Standard block randomisation
Who Masked: Outcomes Assessor
Masking Description: The trial will be single blind for the primary outcome. Devices will be taken off before participants have Doppler imaging at 7 days and 14 days. Data on VTE will be taken by a blinded researcher using information available on hospital information systems.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- geko™ T-3 interventional (Experimental): The geko™ device will be applied bilaterally as soon as possible after randomisation and each geko™ device will be used to deliver one 24-hour dose. Devices will be worn continuously and changed every 24 hours. Treatment will be continued for a maximum of 30 days or until patient recovers mobility, or is discharged into the community, or meet other defined criteria, whichever comes earlier.
  Interventions: Device: geko™ device
- Intermittent Pneumatic Compression (IPC) (No Intervention): Control treatment will be IPC using NHS approved devices as used for standard clinical care. They will be applied to both legs as soon as possible after randomisation. They will not be changed unless damaged or soiled. Treatment will be continued for a maximum of 30 days or until patient recovers mobility, or is discharged into the community, or meet other defined criteria, whichever comes earlier.

INTERVENTIONS:
Device: geko™ device — Neuromuscular electrical stimulation of the peroneal nerve
  Other Names: geko; NMES
  Arms: geko™ T-3 interventional

SUMMARY:
This multicentre, randomised geko™ venous thromboembolism (VTE) prevention study will prospectively collect clinical data on VTE occurrences in immobile patients after stroke, who will be randomised, on a 1:1 allocation, to receive either standard of care (Intermittent Pneumatic Compression) or geko™ neuromuscular electrostimulation device. The aim is to assess the prevention of VTE during a follow-up period of 90 days (three months) post-randomisation.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is a disabling and potentially fatal outcome that may be acquired after having a stroke. The standard treatment to prevent the development of VTE is to give anticoagulation medication. However, this is not recommended in the UK after stroke. Instead the recommended treatment is Intermittent Pneumatic Compression (IPC), where cuffs placed around the lower legs are filled with air to help squeeze the legs and induce blood flow. However, not all patients are able to receive or tolerate IPC treatment. Another treatment which has shown promising results to prevent VTE in immobile patients after stroke, is with a medical device called the geko™ device. The geko™ device is a CE marked medical device which means the manufacturer has checked that the device complies with the essential safety and performance requirements for its' intended use which is to increase blood circulation to help prevent VTE. The aim of this study is to determine if the geko™ device is more effective at preventing VTE in immobile acute stroke patients, than the current IPC standard of care treatment. Following the consent process, stroke patients will be randomised to receive either IPC or geko device. Both devices will be applied until the patient can walk again without help, or for a maximum of 30 days. A compression Doppler exam of the legs will be conducted after 7 days or at discharge if the patient recovers earlier (optional) and after 14 days (mandatory). At 14 days post-randomisation, a patient questionnaire about the comfort of the device, as well as additional health information will be collected. At 30 days after randomisation, additional information about symptomatic DVTs or PEs etc., will be collected from the participant's medical notes. A final follow-up will then be conducted over the phone after 90 days to find out about the patient's recovery, health, mobility and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Clinical diagnosis of acute stroke (WHO criteria)
3. Within 36 hours of symptom onset
4. Not able to get up from a chair/out of bed and walk to the toilet without the help of another person

Exclusion Criteria:

1. Inability to gain consent from the patient, or a declaration from a Personal Consultee or Nominated Consultee
2. Unwitnessed onset with a long lie on the floor before admission
3. Clinically apparent deep vein thrombosis at screening
4. Patient is expected to require palliative care within 14 days
5. Patient does not live in the local catchment area and is expected to be transferred to their local hospital for on-going care.
6. Patient has recently been involved in or is currently involved in a clinical trial for either a medical device or medicinal product, within the past 3 months, with the exception: if co-enrolment is not considered to impact adverse events or outcomes in the opinion of the Chief Investigator. (A live document containing a list of approved studies will be included in a reference document made available to all study sites and available upon request)
7. Contraindications for the use of the geko™ device:

   * Allergy to hydrogel constituents
8. Contraindications to IPC:

   * Severe peripheral vascular disease
   * Large leg ulcers requiring extensive bandaging (small ulcers or skin breaks with flat coverings are not an exclusion)
   * Severe oedema
   * Leg deformities making appropriate fitting impossible
9. Uncontrolled congestive cardiac failure
10. Pregnancy
11. Single or double leg amputations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of any symptomatic or asymptomatic Deep Vein Thrombosis (DVT) in the calf, popliteal or femoral veins or any Pulmonary Embolism (PE). | From randomisation to 30 days. Compression Dopplers at 7 d (optional) and 14 d after randomisation.
  Determine the number of patients diagnosed to have a VTE (DVT and PE), comparing the two groups: geko™ device compared to IPC standard of care. Asymptomatic DVT will be diagnosed using above knee compression Doppler (Compression Duplex Ultrasound) and PE will be diagnosed using ventilation perfusion scan or by computer tomography pulmonary angiogram (CTPA). Compression Dopplers will be conducted any time there is a clinical suspicion of DVT. Above knee compression Dopplers will be conducted at 7 days and 14 days after randomisation, or at patient discharge if patient recovers earlier than 7 d and 14 days post-randomisation.

SECONDARY OUTCOMES:
Device Acceptability | At 14 days after randomisation
  To assess patient tolerability of the geko™ device compared to IPC standard of care, a device acceptability questionnaire will be utilised, which includes questions on discomfort, sleep quality, number of times the device is checked and not in place/not working effectively and number of days the device was worn. Answers to each question will be summarised.
Device effectiveness | At 30 days after randomisation
  Determine frequency of patient death for any cause, confirmed fatal or non-fatal PE, any (symptomatic or asymptomatic) above knee DVT, any (symptomatic or asymptomatic) popliteal or femoral vein DVT or symptomatic calf vein DVT, and combination of these outcomes. The frequency will be compared between the two groups: geko™ device compared to IPC standard of care.
Leg pain level using a Numerical Rating Scale (NRS) score | At 90 days after randomisation
  Assessing pain levels using a Numerical Rating Scale (NRS) score: a line from 0 - 10, where 0 means no pain and 10 is the worst possible pain.
Disability using the modified Rankin score | At 90 days after randomisation
  The modified Rankin score will be used to measure Neurologic Disability. This is a 7-level, clinician reported measure of global disability with possible scores ranging from 0 to 6, where 0 represents "no symptoms at all", 5 represents "severe disability; bedridden, incontinent and requiring constant nursing care and attention" and 6 indicates patient death.
Health related quality of life using EQ-5D-5L | At 90 days after randomisation
  A validated patient reported outcome measure, the first part of the EQ-5D-5L score is a simple 5-level questionnaire: patient mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each question has five response levels from no problems (Level 1) to extreme problems (Level 5). The second part of the EQ-5D is an EQ VAS to record the patient's self-rated health scored on a 0 - 100 scale representing "the worst…" and "the best health you can imagine", respectively.
Patient survival | At 90 days after randomisation
  Death from any cause will be recorded, comparing the two groups: geko™ device compared to IPC standard of care.
Assessment of any symptomatic or asymptomatic DVT or PE | At 90 days after randomisation
  Determine the frequency of VTE (DVT and PE), comparing the two groups: geko™ device compared to IPC standard of care.
Adverse Event Assessments | Up to 30 days after randomisation or discharge, whichever comes earlier
  Incidence of Adverse Events in each group will be recorded.
NIH Stroke Scale/Score (NIHSS) | At 7 days (optional/if practical) and 14 days after randomisation
  The NIHSS scores areas such as level of consciousness, vision, sensation, movement, speech and language with a minimum score of 0 representing no stroke, and 21-42 points representing severe stroke. NIHSS will be compared between the two groups: geko™ device compared to IPC standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Roffe, MD FRCP FESO, Principal Investigator — Keele University, University Hospitals of North Midlands NHS Trust
Locations (18):
- United Kingdom (18):
  - West Suffolk Hospital, Bury St Edmunds, Suffolk
  - Royal United Hospital, Bath
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - The Royal Bournemouth Hospital, Bournemouth
  - Fairfield General Hospital, Bury
  - Addenbrooke's Hospital, Cambridge
  - Kent and Canterbury Hospital, Canterbury
  - Countess of Chester Hospital, Chester
  - Whiston Hospital, Liverpool
  - Northwick Park Hospital, London
  - King's College Hospital, London
  - Milton Keynes University Hospital, Milton Keynes
  - Queen's Medical Centre, Nottingham
  - Salford Royal Hospital, Salford
  - Stepping Hill Hospital, Stockport
  - Royal Stoke University Hospital, Stoke-on-Trent
  - New Cross Hospital, Wolverhampton
  - Yeovil Hospital, Yeovil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Device official website — http://www.gekodevices.com/en-uk/
- See also: Prof Roffe, official website — http://www.stroke-in-stoke.info/the-geko-vte-prevention-study